CLINICAL TRIAL: NCT06765486
Title: Exercise-Induced Hypoalgesia Differences at Proximal and Distal Regions After Applying a Lower Limb Resistance Training or an Upper Limb Resistance Training Protocol: A Randomized Controlled Trial in Healthy Participants
Brief Title: Exercise-Induced Hypoalgesia Differences Between Upper and Lower Limbs Resistance Training Interventions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Álvaro Reina Varona, Principal Investigator, Centro Universitario La Salle
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSEULS-PI-013
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Local Hypoalgesia; Distal Hypoalgesia; Resistance Training; Pressure Pain Thresholds

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lower limb resistance training (Experimental): The participants in the lower limb resistance training group will undergo 3 sets of 5 repetitions of leg extensions with the 5-resistance maximum (5RM), comprising a 5-minute warm-up in cycle ergometer at 1 watt per kg and 60-80 revolutions per minute and 1 set of 5 repetitions with the 10-resistance maximum (10RM).
  Interventions: Other: Lower limb resistance training
- Upper limb resistance training (Experimental): The participants in the upper limb resistance training group will undergo 3 sets of 5 repetitions of brachial biceps curl with the 5RM, comprising a 5-minute warm-up in cycle ergometer at 1 watt per kg and 60-80 revolutions per minute and 1 set of 5 repetitions with the 10RM.
  Interventions: Other: Upper limb resistance training
- Control (No Intervention): Participants in the control group will remain seated for the entire duration of the experiment without receiving any form of distraction.

INTERVENTIONS:
Other: Lower limb resistance training — Exercise intervention with leg extensions on the dominant quadriceps, doing 3 sets of 5 repetitions with the 5RM after a 5-minute warm-up with a cycle ergometer at 1 watt per kg and 60-80 revolutions per minute and 1 set of 5 repetitions with the 10RM. Previously, 72 hours before, the 5RM would have been calculated progressively approaching in sets of 5 repetitions, starting with the lower weight and stopping the test when obtaining an unsuccessful trial (the participant could not manage to lift the weight five times). The previous successful set would be established as the 5RM.
  Arms: Lower limb resistance training
Other: Upper limb resistance training — Exercise intervention with brachial biceps curl on the dominant brachial biceps, doing 3 sets of 5 repetitions with the 5RM after a 5-minute warm-up with a cycle ergometer at 1 watt per kg and 60-80 revolutions per minute and 1 set of 5 repetitions with the 10RM. Previously, 72 hours before, the 5RM would have been calculated progressively approaching in sets of 5 repetitions, starting with the lower weight and stopping the test when obtaining an unsuccessful trial (the participant could not manage to lift the weight five times). The previous successful set would be established as the 5RM.
  Arms: Upper limb resistance training

SUMMARY:
This randomized controlled trial with healthy subjects aims to compare exercise-induced hypoalgesia among three groups: one utilizing a lower limb resistance training intervention, another using an upper limb resistance training, and a control group. The exercise protocol involves 3 sets of 5 repetitions of resistance exercises (brachial biceps curl and leg extensions). Exercise-induced hypoalgesia will be assessed by measuring pressure pain thresholds in the thigh and elbow, comparing exercise interventions with the control group. Additionally, a secondary objective is to compare the lower limb and upper limb resistance training groups in terms of their effects on pressure pain thresholds in the thigh and elbow. Thus, the study anticipates observing differences in local and distal hypoalgesia based on the trained region.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic subjects aged between 18 and 64 years.

Exclusion Criteria:

* Cardiovascular, respiratory, metabolic, neurological, or osteomuscular signs or pathologies.
* History of epilepsy.
* Pregnant.
* Participants who present any type of pain on the day of the measurements or who have frequently suffered pain during the previous 12 weeks.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain pressure threshold (PPT) on dominant quadriceps and dominant brachial biceps | before, immediately after intervention, and 30 minutes after intervention.
  PPT is tested on the muscle belly of the quadriceps on the dominant side, at half of the distance between the anterior-superior iliac spine and the superior pole of the patella, and on the muscle belly of the brachial biceps on the dominant side, at a point one-fourth of the distance from the elbow crease to the lateral border of the acromion. The region to be pressed is marked with a pen. The patient is instructed to report the first appearance of the sensation of "discomfort". An ascending ramp of 0.5 kg/cm/s is applied, at the rhythm of a metronome. The instrument measures 0 to 25 kg, with a higher score interpreted as a hypoalgesia response. The measurement is started on the quadriceps and alternated with the biceps until 3 measurements of each region are obtained. Each measurement in the same region is obtained after 30 seconds of rest. This protocol has demonstrated high inter-observer reliability measuring healthy subjects (ICC = 0.91).

SECONDARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) | before intervention (up 5 minutes)
  7-item questionnaire on the level of physical activity at different intensities (high, moderate, and low) and hours sitting.
  A higher score means higher weekly physical activity
Physical Activity Readiness Questionnaire (PAR-Q) | before intervention (up 5 minutes)
  7-item questionnaire that assesses an individual's readiness to engage in physical activity based on whether any known contraindications have been ruled out by the participant.
  If all the questions are negative, the participant can safely engage in a physical activity.
Fatigue Assessment Scale (FAS) | before intervention (up 5 minutes)
  10-item questionnaire that allows for the evaluation of the participant's current level of fatigue. This instrument measures 10 to 50 points.
  A higher score means higher fatigue.
Rate of perceived exertion (RPE) | immediately after intervention (up 10 seconds)
  RPE Borg CR-10 is used to measure how hard your body works during physical activity. It runs from 0 - 10, using numbers to rate how much effort an activity takes. Higher scores indicate a higher perception of effort.

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU LaSalle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No